CLINICAL TRIAL: NCT05626439
Title: An Open-Label, Randomized, Single-Dose, 2-Way Crossover Study to Evaluate The Relative Bioavailability of Staccato Alprazolam Compared to Oral Alprazolam in Healthy Study Participants
Brief Title: A Relative Bioavailability Study of Staccato Alprazolam Versus Oral Alprazolam in Healthy Study Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UP0104
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Bioavailability; Phase 1; Staccato alprazolam
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Sequence AB (Experimental): Study participants randomized into this arm will receive single dose of Staccato alprazolam followed by single dose of oral alprazolam at pre-specified time points in the sequence AB.
  Interventions: Drug: Staccato alprazolam; Drug: Oral alprazolam
- Treatment Sequence BA (Experimental): Study participants randomized into this arm will receive single dose of oral alprazolam followed by single dose of Staccato alprazolam at pre-specified time points in the sequence BA.
  Interventions: Drug: Staccato alprazolam; Drug: Oral alprazolam

INTERVENTIONS:
Drug: Staccato alprazolam — Study participants will receive single dose of Staccato alprazolam by inhalation at pre-specified time points.
  Other Names: UCB7538
Drug: Oral alprazolam — Study participants will receive single dose of oral alprazolam at pre-specified time points.
  Other Names: Xanax

SUMMARY:
The purpose of the study is to evaluate the relative bioavailability of alprazolam in plasma following a single dose of Staccato alprazolam compared to a single dose of oral alprazolam under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring, at the Screening Visit or on Day -1 of the first Treatment Period
* Participant has a body weight of at least 45 kg (female) and 50 kg (male) and body mass index (BMI) within the range 18 to 35 kg/m^2 (inclusive) at the Screening Visit or on Day -1 of the first Treatment Period
* Participants may be male or female:

A male participant must agree to use contraception as detailed in the protocol during the Treatment Periods and for at least 7 days after the second Investigational Medicinal Product (IMP) administration and must refrain from donating sperm during this period.

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

* Not a woman of childbearing potential (WOCBP) as defined in the protocol OR A WOCBP who agrees to follow the contraceptive guidance in the protocol during the Treatment Periods and for at least 30 days after the second IMP administration

Exclusion Criteria:

* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Participant has a history or present condition of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological, cerebrovascular, or other major disorders capable of significantly altering the absorption, metabolism, or elimination of Investigational Medicinal Product (IMP); constituting a risk when taking the IMP; or interfering with the interpretation of data
* Participant has abnormal blood pressure (BP) or heart rate (HR) at the Screening Visit or on Day -1 of the first Treatment Period (as stated in the protocol). Study participants must have BP and HR within normal range in the supine position after 5 minutes of rest (systolic BP [SBP]: 90 mmHg to 140 mmHg, diastolic BP [DBP]: 50 mmHg to 90 mmHg, HR: 50 beats per minute to 100 beats per minute (bpm). In case of an out-of-range result, 1 repeat will be allowed. If the readings are out of range again, the study participant will not be included
* Participant has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt) or has had suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Screening/Baseline" version of the Columbia Suicide Severity Rating Scale (C-SSRS) at the Screening Visit
* Participant has had a positive test for Severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) or clinical signs/symptoms consistent with coronavirus disease 2019 (COVID-19) such as fever, persistent cough, shortness of breath, fatigue, and loss or change to senses of smell or taste during the 4 weeks prior to the Screening Visit or Day -1 of the first Treatment Period
* Participant has a condition for which oral alprazolam is contraindicated (eg, myasthenia gravis, severe respiratory insufficiency, sleep apnea syndrome, and severe hepatic insufficiency)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to infinity (AUC) of alprazolam | Plasma samples will be collected from Baseline (Day 1 predose) at predefined time points (up to Day 3)
  AUC = Area under the plasma concentration-time curve from time zero to infinity
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-t)) of alprazolam | Plasma samples will be collected from Baseline (Day 1 predose) at predefined time points (up to Day 3)
  AUC(0-t) = Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration
Maximum plasma concentration (Cmax) of alprazolam | Plasma samples will be collected from Baseline (Day 1 predose) at predefined time points (up to Day 3)
  Cmax = Maximum plasma concentration

SECONDARY OUTCOMES:
Percentage of study participants with treatment-emergent adverse events (TEAEs) | From Baseline (Day 1) of Treatment Period 1 to the end of Safety Follow-Up (up to 25 days)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication.
Percentage of study participants with serious treatment-emergent adverse events (serious TEAEs) | From Baseline (Day 1) of Treatment Period 1 to the end of Safety Follow-Up (up to 25 days)
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  Results in death Is life-threatening Requires inpatient hospitalization or prolongation of existing hospitalization Results in persistent disability/incapacity Is a congenital anomaly/birth defect Important medical events referred to in the Protocol.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0104 1001, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.